CLINICAL TRIAL: NCT02198287
Title: A Single Increasing Dose Safety and Tolerability Study (Dose Extension) After Inhalational Administration of BIIX 1 XX (Single Doses: 800 - 2000 mcg) in Healthy Young Male Volunteers (Randomised, Double-blind, Placebo-controlled)
Brief Title: Dose Extension Study of BIIX 1 XX in Healthy Young Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1150.7
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BIIX 1 XX, rising doses (Experimental)
  Interventions: Drug: BIIX 1 XX inhalation solution
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIX 1 XX inhalation solution — single doses of 800, 1000, 1200, 1400, 1600, 1800, or 2000 mcg
  Arms: BIIX 1 XX, rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
Safety, tolerability and pharmacokinetic study of BIIX 1 XX in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, based on a complete medical examination
* Age range from 21 to 50 years
* Participant must be within +/- 20 % of their normal weight (Broca-Index)
* Participant must provide written informed consent

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) or laboratory tests deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (≥ 24 hours) within at least one month or less than then half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial within seven days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to start of the study
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse
* Drug abuse
* Blood donation (> 100 ml) within four weeks prior to administration
* Other disease or abnormality of clinical relevance
* Excessive physical activities within two weeks prior to administration or during the trial

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 1999-01; Primary Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 22 days
Number of patients with clinically relevant changes in vital parameters (Blood pressure, Pulse rate) | up to 8 days after drug administration
Number of patients with clinically relevant changes in electrocardiogram (ECG) | up to 8 days after drug administration
Number of patients with clinically relevant changes in impedance cardiography | pre-dose, 10 and 30 minutes after administration
Number of patients with clinically relevant changes in cutaneous microcirculation | pre-dose, 10 and 30 minutes after administration
Number of patients with clinically relevant changes in safety laboratory parameters | up to 8 days after drug administration

SECONDARY OUTCOMES:
Maximum concentration of the drug in plasma (Cmax) | up to 168 hours after drug administration
Area under the plasma drug concentration-time curve from zero time to the last time point of measurement (AUC0-tz) | up to 168 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | up to 168 hours after drug administration
Clearance, divided by f (CL/f) | up to 168 hours after drug administration